CLINICAL TRIAL: NCT03602742
Title: Comparison of 24-hour Holter Monitoring Versus 14-day Continuous ECG Patch Monitoring EZYPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sigknow Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SIGEZYZ20170828
Record Dates: First submitted 2018-05-24; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Atrial Fibrillation; Arrhythmias, Cardiac
Keywords: Atrial Fibrillation; Arrhythmias, Cardiac; EZYPRO ECG Recorder; ECG monitor; Long term ECG monitor; 14-day ECG monitor
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 24-hour Holter and 14-day EZYPRO® (Other): This is an open-label study to investigate the functional features of prolonged monitoring by 14-day EZYPRO® to improve the medical care and/or diagnosis for the patient with arrhythmia. One arm included.
  Interventions: Device: EZYPRO®

INTERVENTIONS:
Device: EZYPRO® — Wear two devices including 24-hour Holter and 14-day continuous EZYPRO® to evaluate the performance
  Other Names: 24-hour Holter

SUMMARY:
This is an open-label study to investigate the functional features of prolonged monitoring by 14-day EZYPRO® to improve the medical care and/or diagnosis for the patient with arrhythmia. Patients will be enrolled by outpatient basis from two clinical study sites. Enrolled patients will wear a traditional 24-hour Holter monitor and an 14-day EZYPRO® which can provide monitoring data for up to 14 days. This study will allow a direct comparison between two devices.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent before enrollment into the study
* Are able to communicate with the investigators
* With suspected arrhythmia related signs and symptoms, judged by the investigators
* Patients intend to wear ECG moniotrs
* Males and females, 20 years of age or older

Exclusion Criteria:

* Patients with skin allergies or injury, judged by investigators
* Patients with specific arrhythmia or specific treatments, interfere with study evaluations, judged by investigators
* Pregnant women
* Currently participating in another trial or who participated in a previous clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare the detection difference of any type of arrhythmia between 14-day continuous ECG patch and 24-hour Holter monitor device among patients with suspected cardiac arrhythmia events over total wearing time | Up to14 days
  The arrhythmia events of 14-day continuous ECG patch monitor (investigational device) and 24-hour Holter monitor will be analyzed by the qualified ECG technicians and determined by physician investigators at the study sites. Arrhythmia events are defined as detection of any 1 of 6 arrhythmias, including:
  * Supraventricular tachycardia (>4 beats, not including atrial fibrillation or flutter)
  * Atrial fibrillation/flutter (>4 beats)
  * Pause >3 seconds
  * Atrioventricular block (Second-degree, 2:1 or third-degree atrioventricular block, need an advanced determination by the investigators)
  * Ventricular tachycardia (>4 beats)
  * Polymorphic ventricular tachycardia/ventricular fibrillation In the end, all the detection will be confirmed by the investigators.
  McNemar's tests will be used to compare the matched pairs of proportion data.

SECONDARY OUTCOMES:
The wearing time of 14-day continuous ECG patch (Study Compliance) | Up to14 days
  The wearing time will be recorded as the day of 14-day continuous ECG patch removal after stating monitoring. Kaplan-Meier method will be reported for total wearing time. The mean value along with two-sided 95% confidence intervals will be report as well.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shien Wen, Principal Investigator — Chang Gung Medical Foundation, Linkou; Shih-Lin Chang, Principal Investigator — Veterans General Hospital
Locations (2):
- Taiwan (2):
  - Taipei Veterans General Hospital, Taiwan, Taipei
  - Chang Gung Medical Foundation, Linkou, Taoyuan District